CLINICAL TRIAL: NCT02810795
Title: Dynamic Stress Perfusion ct for Detection of Inducible Myocardial Ischemia
Acronym: SPECIFIC
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University Hospital Tuebingen (Other); Siemens Medical Solutions (Industry); Bayer (Industry); University of Erlangen-Nürnberg (Other); University Medical Center Groningen (Other); Mie University (Other); University Hospital, Zürich (Other); Queen Mary University of London (Other); University Hospital Munich (Other)
Responsible Party: Principal Investigator, Trialbureau radiology, Dr. K. Nieman MD, PHD, Erasmus Medical Center
Other Study IDs: SPECIFIC
Record Dates: First submitted 2016-06-07; First posted 2016-06-23 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary; Artery; Computed tomography; FFR; CT myocardial perfusion; Dynamic
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Diagnostic detection of coronary artery disease — Myocardial perfusion defect on dynamic CT perfusion imaging, and diagnostic accuracy as compared invasive FFR.

SUMMARY:
The purpose of this study is to determine the diagnostic accuracy of MPICT for the detection of hemodynamically relevant coronary stenosis (as determined by invasive FFR) in patients with suspected or known CAD clinically referred for invasive angiography.

DETAILED DESCRIPTION:
Rationale: Cardiac computed tomography (CT) provides accurate assessment of the coronary arteries and detects significant coronary stenosis with high diagnostic accuracy. However, the hemodynamic relevance of these stenotic lesion remains unclear, although highly relevant for clinical decision-making. Recent technical developments with third-generation dual-source CT allow to determine myocardial perfusion during hyperemia and thus for assessment of the hemodynamic relevance of coronary lesions using a dynamic acquisition mode. To date, there is only very limited evidence of the feasibility of this approach stemming from single-center studies with varying standards of reference.

Objective: To determine the diagnostic accuracy of MPICT for the detection of hemodynamically relevant coronary stenosis (as determined by invasive FFR) in patients with suspected or known CAD clinically referred for invasive angiography. In an optional sub-study the diagnostic accuracy of MPICT for the detection of myocardial perfusion defects as determined by cardiac magnetic resonance imaging (CMRI) will be investigated.

Study design: Observational cohort study with fractional flow reserve (FFR) during invasive angiography as the reference standard.

Study population: Patients with known or suspected CAD clinically referred for invasive angiography.

Main study parameters: Myocardial perfusion defect on dynamic CT perfusion imaging, and diagnostic accuracy as compared invasive FFR.

Co Principle Investigators Koen Nieman MD PhD, Erasmus University Medical Center Fabian Bamberg MD PhD, University of Tübingen.

Investigators Valerie Schmidt-Honndorf PhD, University of Tübingen Tobias Geisler MD PhD, University of Tübingen Joost Daemen MD PhD, Erasmus University Medical Center Adriaan Coenen MD, Erasmus University Medical Center Stephan Achenbach MD PhD, Erlangen University Micheala M. Hell MD, Erlangen University Rozemarijn Vliegenthart MD PhD, UMC Groningen Pim van der Harst MD PhD, UMC Groningen Francesca Pugliese MD PhD, Queen Mary University of London Kakuya Kitagawa MD PhD, Mie University Hatem Alkadhi MD PhD, University Hospital Zurich, Switzerland Robert Manka MD PhD, University Hospital Zurich, Switzerland

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75 years
* Stable angina symptoms, suspected or known CAD, and referred for invasive angiography on clinical grounds.
* Ability to provide informed consent
* Ability to perform a 20-30 second breath hold

Exclusion Criteria:

* Hemodynamically and clinically unstable condition (angina at rest, malignant arrhythmias)
* Prior, documented myocardial infarction, other than (procedure related) minor type II myocardial infarction, which includes Q waves on the ECG or evidence of myocardial infarction on prior non-invasive imaging.
* Prior stenting or coronary artery bypass graft surgery
* Significant other cardiovascular conditions affecting the interpretation of MPICT, including, but not limited to: clinical heart failure, IECD (pacemaker/ICD), severe valvular heart disease or prosthetic valves, significant intra-cardiac shunting or other relevant congenital heart disease.
* eGFR<60 ml/kg/min
* BMI>30 kg/m2, or weight >120 kg.
* Atrial fibrillation or other arrhythmia, >6 ectopic beats / min
* Known or suspected allergy to iodinated contrast medium
* Pregnancy cannot be excluded
* Contra-indications for adenosine: bronchial asthma, second or third degree atrioventricular block, blood pressure <110/70 mmHg, allergies or severe side effects in the past.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with know or suspect coronary artery diseased, referred for invasive coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Myocardial perfusion | For each patient within 4 weeks of the CT perfusion acquisition
  invasive fractional flow reserve measurement

SECONDARY OUTCOMES:
Presence of myocardial perfusion defect on MPIMRI | For each patient within 1 week before invasive fractional flow reserve measurement
Per patient assessment of hemodynamically significant CAD | For each patient within 4 weeks of the CT perfusion acquisition
Ischemia per standardized myocardial segment | For each patient within 4 weeks of the CT perfusion acquisition
Coronary stenosis by CTA per territory (branch) | For each patient within 4 weeks of the CT perfusion acquisition
Coronary stenosis by invasive angiography per territory (branch) | For each patient within 4 weeks of the CT perfusion acquisition
Demographics. | For each patient within 1 week before invasive fractional flow reserve measurement
Cardiovascular risk factors | For each patient within 1 week before invasive fractional flow reserve measurement
'Image quality, based on the DICOM images measured by experienced readers." | Through study completion, an average of 1 to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Koen Nieman, MD PHD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soschynski M, Storelli R, Birkemeyer C, Hagar MT, Faby S, Schwemmer C, Nous FMA, Pugliese F, Vliegenthart R, Schlett CL, Nikolaou K, Krumm P, Nieman K, Bamberg F, Artzner CP. CT Myocardial Perfusion and CT-FFR versus Invasive FFR for Hemodynamic Relevance of Coronary Artery Disease. Radiology. 2024 Aug;312(2):e233234. doi: 10.1148/radiol.233234. PMID 39162632
- [Derived] Nous FMA, Geisler T, Kruk MBP, Alkadhi H, Kitagawa K, Vliegenthart R, Hell MM, Hausleiter J, Nguyen PK, Budde RPJ, Nikolaou K, Kepka C, Manka R, Sakuma H, Malik SB, Coenen A, Zijlstra F, Klotz E, van der Harst P, Artzner C, Dedic A, Pugliese F, Bamberg F, Nieman K. Dynamic Myocardial Perfusion CT for the Detection of Hemodynamically Significant Coronary Artery Disease. JACC Cardiovasc Imaging. 2022 Jan;15(1):75-87. doi: 10.1016/j.jcmg.2021.07.021. Epub 2021 Sep 15. PMID 34538630